CLINICAL TRIAL: NCT02038881
Title: Randomized, Open-label Phase II Trial to Assess the Safety and Immunogenicity of MVA-BN Smallpox Vaccine When Increasing the Number of Injections Compared to the Standard Regimen in Immunocompromised Subjects With HIV Infection
Brief Title: Randomized, Open-label Phase II Trial to Assess the Safety and Immunogenicity of MVA-BN Smallpox Vaccine in Immunocompromised Subjects With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-037
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (standard regimen) (Experimental): One injection at Day 0 and Day 28 with IMVAMUNE® (MVA-BN®)
  Interventions: Biological: IMVAMUNE®
- Group 2 (double dose regimen) (Experimental): Two injections at Day 0 and two injections at Day 28 with IMVAMUNE® (MVA-BN®)
  Interventions: Biological: IMVAMUNE®
- Group 3 (booster regimen) (Experimental): One injection at Day 0 and Day 28 and one booster injection at week 12 with IMVAMUNE® (MVA-BN®)
  Interventions: Biological: IMVAMUNE®

INTERVENTIONS:
Biological: IMVAMUNE® — 0.5 ml Modified Vaccinia Ankara Strain - Bavarian Nordic (MVA-BN®) smallpox vaccine containing at least 1 x 10E8 TCID50 per ml
  Other Names: IMVANEX®; MVA-BN® smallpox vaccine

SUMMARY:
The main purpose of this clinical trial is to generate additional safety data in a highly immunocompromised population. HIV-infected persons are considered excellent candidates to represent the highly immunocompromised population for enrolment in this trial. Additionally, the immune system's response (protection against smallpox as measured by the amount of antibodies produced) following injections of MVA-BN® smallpox vaccine will be evaluated. All participants in this trial will be randomly and evenly assigned to one of three groups to receive two, three or four injections. Group 1 will receive the standard regime consisting of one dose at each vaccination time point, Group 2 will receive two doses at each vaccination time point and Group 3 will receive a booster vaccination 12 weeks after the standard vaccination schedule with MVA-BN® smallpox vaccine. Participation in the trial is scheduled to last up to 75 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 18-45 years, vaccinia-naïve.
2. HIV-1 infection documented by ELISA and confirmed by Western blot at any time prior to study entry. HIV-1 deoxyribonucleic acid (DNA) polymerase chain reaction (PCR), HIV-1 culture, HIV-1 antigen, plasma HIV-1 ribonucleic acid (RNA), or a second antibody test other than ELISA is acceptable as an alternative test at any time prior to study entry.
3. On stable antiretroviral therapy (ART) i.e. Combination ART for at least 6 months. Subject must be on the same ART regimen for at least 12 weeks with no change prior to enrollment in this clinical trial.
4. Screening HIV-1 RNA < 200 copies/ml by US Food and Drug Administration (FDA) approved PCR assay within 45 days prior to study entry.
5. Current CD4 counts ≥ 100 cells/µl ≤ 500 cells/µl.
6. Documented nadir CD4 count < 200 cells/µl at any time prior to enrollment.
7. Hemoglobin ≥ 9.0 g/dl for female subjects, ≥ 10.0 g/dl or male subjects.
8. Platelets ≥ 100,000/mm3.
9. Ability and willingness of subject to provide written informed consent.
10. Body Mass Index (BMI) ≥ 18.5 and < 35 kg/m2.
11. Women of childbearing potential (WOCBP) must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the trial, and must avoid becoming pregnant for at least 28 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal (defined as ≥ 12 months without a menstrual period) or surgically sterilized. Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products).
12. WOCBP must have a negative serum pregnancy test at screening (SCR) and a negative urine pregnancy test within 24 hours prior to each vaccination.
13. Absolute neutrophil count cells ≥ 750/mm3.
14. Adequate renal function defined as a calculated Creatinine Clearance (CrCl) > 60 ml/min as estimated by the Cockcroft-Gault equation.

    1. For men: (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dl x 72) = CrCl (ml/min)
    2. For women: multiply the result by 0.85 = CrCl (ml/min).Adequate hepatic function defined as: Total bilirubin ≤ 2 x upper limit normal (ULN) in the absence of other evidence of significant liver disease
15. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 2.5 x ULN.
16. Troponin I < 2 x ULN at entry in the clinical trial.
17. Electrocardiogram (ECG) without clinically significant findings (e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions (PVC) in a row, ST elevation consistent with ischemia).

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Typical vaccinia scar.
3. Known or suspected history of smallpox vaccination.
4. History of vaccination with any poxvirus-based vaccine.
5. Uncontrolled serious infection, i.e. not responding to antimicrobial therapy.
6. History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject or would limit the subject's ability to complete the trial including uncontrolled diabetes as according to the 'Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events' Version 1.0, December 2004, Clarification August 2009.
7. History of or active autoimmune disease, persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
8. Known or suspected impairment of immunologic function except those defined in the inclusion criteria, including, but not limited to clinically significant liver disease, diabetes mellitus type I and moderate to severe kidney impairment.
9. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site.
10. History or clinical manifestation of clinically significant and severe hematological, pulmonary, central nervous, cardiovascular or gastrointestinal disorders (except HIV infection, chronic or active Hepatitis-B-Virus or Hepatitis-C-Virus infection).
11. Clinically significant psychiatric disorder not adequately controlled by medical treatment.
12. History of coronary heart disease, myocardial infarction, angina pectoris, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
13. Known history of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before age 50 years.
14. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof). NOTE: This criterion applies only to subjects 20 years of age and older.
15. Current alcohol abuse (40 g/day for at least 6 month) and/or intravenous and/or intranasal drug abuse (within the past 6 months).
16. Known allergy to MVA-BN® vaccine or any of its constituents, e.g. tris (hydroxymethyl)-amino methane, including known allergy to egg or aminoglycosides.
17. History of anaphylaxis or severe allergic reaction to any vaccine.
18. Acute disease (illness with or without a fever) at the time of enrollment.
19. Body temperature ≥ 100.4°F (≥ 38.0°C) at the time of enrollment.
20. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after trial vaccination.
21. Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior to or after trial vaccination.
22. Use of immunosuppressant or immunomodulatory agents including systemic glucocorticoids (excluding nasal or inhaled steroids), tacrolimus, sirolimus, rapamycin, mycophenolate, cyclosporine, TNF-alpha blockers or antagonists, azathioprine, interferon, growth factors, or intravenous immunoglobulin in the 60 days prior to enrollment in this clinical trial.
23. Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
24. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit.
25. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the first dose of the trial vaccine, or planned administration of such a drug during the trial period.
26. Trial personnel.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar T Overton, MD, Principal Investigator — University of Alabama at Birmingham
Locations (12):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Health for Life Clinic Little Rock, Little Rock, Arkansas
  - Quest Clinical Research, San Francisco, California
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Infectious Disease Associats of NW Florida Center for Prevention and Treatment of Infections Infectious Diseases Associates of NW FL, Pensacola, Florida
  - Rowan Tree Medical, Wilton Manors, Florida
  - University of Illinois - Chicago, Chicago, Illinois
  - University of Iowa Departments of Internal Medicine and Microbiology University of Iowa, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pennsylvania Clinical Trials Unit, Philadelphia, Pennsylvania
- Puerto Rico (2):
  - Clinical Research Puerto Rico, Inc., San Juan, PR
  - Fundacion de Investigacion, San Juan, PR

REFERENCES:
- [Derived] Overton ET, Lawrence SJ, Stapleton JT, Weidenthaler H, Schmidt D, Koenen B, Silbernagl G, Nopora K, Chaplin P. A randomized phase II trial to compare safety and immunogenicity of the MVA-BN smallpox vaccine at various doses in adults with a history of AIDS. Vaccine. 2020 Mar 4;38(11):2600-2607. doi: 10.1016/j.vaccine.2020.01.058. Epub 2020 Feb 11. PMID 32057574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 12 sites in the US
Period: Overall Study
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Started | 27 | 29 | 31
Completed | 24 | 29 | 30
Not Completed | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — incarcerated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen) | Total
Number analyzed (Participants) | 27 | 29 | 31 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.66) | 33.1 (6.67) | 36.6 (5.43) | 35 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 12
  Male | 23 | 24 | 28 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 0
  Oriental/Asian | 0 | 0 | 0 | 0
  Black/African American | 16 | 18 | 16 | 50
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 1 | 1
  White/Caucasian | 10 | 10 | 14 | 34
  Other | 1 | 1 | 0 | 2
  Hispanic or Latino | 5 | 4 | 3 | 12
  Not Hispanic or Latino | 22 | 25 | 28 | 75
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 31 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SAEs
Description: Occurrence, relationship and intensity of any serious AE (SAE)
Time Frame: within 75 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
Participants
  Any SAE | 0 | 0 | 2
  Any SAE with intensity >= Grade 3 | 0 | 0 | 2
  Any SAE assessed as related to vaccine | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With AESIs
Description: Occurrence, relationship to the trial vaccine, and intensity of any adverse event of special interest (AESI)
Time Frame: within 75 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
Participants
  Any AESI | 0 | 0 | 1
  Any AESI with intensity >= Grade 3 | 0 | 0 | 0
  Any AESI assessed as related to vaccine | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Related Grade >=3 Adverse Events
Description: Number of Participants with any Grade >=3 Adverse Event probably, possibly, or definitely related to the study vaccine. Pooled solicited and unsolicited AEs.
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
Participants | 4 | 5 | 3

4. Secondary Outcome: Number of Unsolicited Non-serious Adverse Events: Relationship to Vaccination
Description: Occurrence of unsolicited non-serious AEs by relationship to study vaccine
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Number; unit: events
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
events
  Unrelated/None | 4 | 4 | 13
  Unlikely | 1 | 2 | 1
  Possible | 1 | 1 | 0
  Probable | 0 | 0 | 1
  Definite | 0 | 0 | 0

5. Secondary Outcome: Number of Unsolicited Non-serious Adverse Events: Intensity
Description: Occurrence of unsolicited non-serious AEs by Intensity
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Number; unit: events
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
events
  Mild | 4 | 7 | 9
  Moderate | 1 | 0 | 6
  Severe | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Number of participants with solicited local AEs (redness, swelling, induration, pruritus, and pain) by intensity. Percentages based on subjects with at least one completed diary card. [Injection site erythema, injection site swelling and injection site induration--all sizes measured in diameter with max severity of: 0=0, 1 = <30 mm, 2 = ≥30 - <100 mm, 3 = ≥100 mm. Injection site pruritus: 0=absent, 1=mild, 2=moderate, 3=severe. Injection site pain: 0=absent, 1=painful to touch, 2=painful when limb is moved, 3=spontaneously painful/prevents normal activity.]
Time Frame: within 8 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
Participants
  Injection Site Pain, Grade 1 | 5 | 4 | 11
  Injection Site Pain, Grade 2 | 10 | 11 | 10
  Injection Site Pain, Grade 3 | 2 | 4 | 1
  Injection Site Erythema, Grade 1 | 7 | 11 | 15
  Injection Site Erythema, Grade 2 | 1 | 0 | 3
  Injection Site Erythema, Grade 3 | 0 | 0 | 0
  Injection Site Swelling, Grade 1 | 9 | 9 | 9
  Injection Site Swelling, Grade 2 | 1 | 1 | 4
  Injection Site Swelling, Grade 3 | 0 | 0 | 0
  Injection Site Induration, Grade 1 | 7 | 5 | 9
  Injection Site Induration, Grade 2 | 1 | 1 | 1
  Injection Site Induration, Grade 3 | 0 | 0 | 0
  Injection Site Pruritus, Grade 1 | 7 | 6 | 15
  Injection Site Pruritus, Grade 2 | 4 | 2 | 3
  Injection Site Pruritus, Grade 3 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Solicited General AEs
Description: Number of Participants with solicited systemic/general AEs (pyrexia, headache, myalgia, nausea, fatigue, and chills) by intensity. Percentages based on subjects with at least one completed diary card. [Body temperature: 0 = <99.5 F (<37.5 C), 1 = ≥99.5 - <100.4 F (≥37.5 - <38.0 C), 2= ≥100.4 - <102.2 F (≥38.0 - <39.0 C), 3= ≥102.2 - <104.0 F (≥39.0 - <40.0 C), 4= ≥ 104.0 F (≥40.0 C); pyrexia is defined as oral temperature ≥ 100.4 F (≥ 38.0 C).] [Headache, myalgia, nausea, chills and fatigue: 0 = none, 1 = mild: easily tolerated, minimal discomfort and no interference with daily activity, 2 = moderate: some interference with daily activity, 3 = severe: prevents daily activity.]
Time Frame: within 8 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
Participants
  Pyrexia, Grade 1 | 0 | 0 | 0
  Pyrexia, Grade 2 | 1 | 0 | 0
  Pyrexia, Grade 3 | 0 | 0 | 0
  Headache, Grade 1 | 8 | 5 | 6
  Headache, Grade 2 | 1 | 3 | 3
  Headache, Grade 3 | 0 | 2 | 1
  Myalgia, Grade 1 | 6 | 6 | 8
  Myalgia, Grade 2 | 2 | 6 | 4
  Myalgia, Grade 3 | 1 | 0 | 1
  Chills, Grade 1 | 4 | 4 | 5
  Chills, Grade 2 | 2 | 2 | 1
  Chills, Grade 3 | 1 | 0 | 0
  Nausea, Grade 1 | 3 | 4 | 4
  Nausea, Grade 2 | 3 | 0 | 2
  Nausea, Grade 3 | 0 | 2 | 0
  Fatigue, Grade 1 | 5 | 4 | 5
  Fatigue, Grade 2 | 2 | 5 | 5
  Fatigue, Grade 3 | 2 | 2 | 1

8. Secondary Outcome: CD4+ T Cell Counts
Description: Mean CD4+ T-cell counts over time
Time Frame: within 15 days after each vaccination
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: CD4 count (cells/µL)
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 27 | 29 | 31
CD4 count (cells/µL)
  Screening | 304.9 (104.77) | 295.3 (111.10) | 349.6 (133.71)
  Week 2 | 337.4 (118.18) | 357.0 (157.87) | 335.7 (111.11)
  Week 6 | 319.1 (117.91) | 365.4 (197.04) | 345.0 (96.22)
  Week 14 | NA (NA) — N/A=week 14 visit not scheduled for Group 1 | NA (NA) — N/A=week 14 visit not scheduled for Group 2 | 351.9 (114.53)

9. Secondary Outcome: Geometric Mean Titers (GMT) Measured by Enzyme-linked Immunosorbent Assay (ELISA) at All Immunogenicity Sampling Points
Description: GMTs based on vaccinia-specific ELISA. Titers below the detection limit are included with a value of '1'.
Time Frame: within 64 weeks
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
Titer
  Week 0 | 1.5 [0.8 to 2.6] | 1.2 [0.8 to 1.7] | 1.8 [0.9 to 3.5]
  Week 4 | 40.0 [15.3 to 105.1] | 47.1 [20.7 to 107.1] | 41.8 [16.2 to 107.8]
  Week 6 | 552.2 [337.1 to 904.4] | 846.1 [475.3 to 1506.1] | 726.1 [371.3 to 1419.8]
  Week 12 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 193.1 [90.9 to 410.5]
  Week 14 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 1591.2 [1158.1 to 2186.3]
  Week 30/38 | 34.6 [12.2 to 98.5] | 30.8 [11.3 to 83.5] | 143.3 [67.6 to 303.9]
  Week 56/64 | 25.2 [8.4 to 75.7] | 27.5 [9.6 to 79.2] | 116.2 [57.9 to 233.2]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 4 = 0.851, 95% CI 2-sided [0.258 to 2.800]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 6 = 0.653, 95% CI 2-sided [0.319 to 1.333]
Statistical Analysis 3: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 30 = 1.126, 95% CI 2-sided [0.291 to 4.352]
Statistical Analysis 4: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 56 = 0.916, 95% CI 2-sided [0.220 to 3.819]
Statistical Analysis 5: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 / Group 1) at Week 4 = 1.045, 95% CI 2-sided [0.292 to 3.741]
Statistical Analysis 6: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 / Group 1) at Week 6 = 1.315, 95% CI 2-sided [0.598 to 2.892]

10. Secondary Outcome: ELISA GMT 2 Weeks Following the Second Vaccination (Group 2 Compared to Group 1 and Group 3 (Combined))
Description: GMTs based on vaccinia-specific ELISA. Titers below the detection limit are included with a value of '1'.
Time Frame: Week 6
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Group 1 and 3 Combined: Pooling of Groups 1 and 3 (same dose/regimen before booster vaccination in Group 3)
- Group 2: Double dose regimen
Arm/Group | Group 1 and 3 Combined | Group 2
Number analyzed (Participants) | 46 | 23
Titer | 644.6 [422.7 to 983.0] | 846.1 [475.3 to 1506.1]
Statistical Analysis 1: Comparison: Group 1 and 3 Combined vs Group 2; Test type: Other; GMT Ratio (Group 1+3 [pooled] / Group 2) = 0.762, 95% CI 2-sided [0.385 to 1.507]

11. Secondary Outcome: ELISA GMT 2 Weeks Following the Last Vaccination
Description: GMTs based on vaccinia-specific ELISA. Titers below the detection limit are included with a value of '1'.
Time Frame: Week 6 (Groups 1 and 2), Week 14 (Group 3)
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
Titer | 552.2 [337.1 to 904.4] | 846.1 [475.3 to 1506.1] | 1591.2 [1158.1 to 2186.3]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 1 [W6]/ Group 3 [W14) = 0.347, 95% CI 2-sided [0.200 to 0.603]
Statistical Analysis 2: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT ratio (Group 2 [W6]/ Group 3 [W14]) = 0.532, 95% CI 2-sided [0.285 to 0.992]

12. Secondary Outcome: ELISA GMT During Follow-up
Description: GMTs based on vaccinia-specific ELISA. Titers below the detection limit are included with a value of '1'. Participants discontinued prior to the follow-up visits are excluded.
Time Frame: Weeks 30 and 56 (Groups 1 and 2), Weeks 38 and 64 (Group 3)
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 18 | 22 | 24
Titer
  Week 30/38 | 34.6 [12.2 to 98.5] | 30.8 [11.3 to 83.5] | 143.3 [67.6 to 303.9]
  Week 56/64 | 25.2 [8.4 to 75.7] | 27.5 [9.6 to 79.2] | 116.2 [57.9 to 233.2]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 [W38]/ Group 1 [W30]) = 4.138, 95% CI 2-sided [1.241 to 13.793]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 [W64]/ Group 1 [W56]) = 4.608, 95% CI 2-sided [1.365 to 15.558]
Statistical Analysis 3: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 2 [W30]/ Group 3 [W38]) = 0.215, 95% CI 2-sided [0.066 to 0.699]
Statistical Analysis 4: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 2 [W56]/ Group 3 [W64]) = 0.237, 95% CI 2-sided [0.072 to 0.782]

13. Secondary Outcome: GMTs Measured by Plaque Reduction Neutralization Test (PRNT) at All Immunogenicity Sampling Points
Description: GMTs based on vaccinia-specific PRNT. Titers below the detection limit are included with a value of '1'.
Time Frame: within 64 weeks
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
Titer
  Week 0 | NA [NA to NA] — None of the participants have titer values above the detection limit. | NA [NA to NA] — None of the participants have titer values above the detection limit. | 1.2 [0.8 to 1.9]
  Week 4 | 3.9 [1.9 to 8.1] | 4.8 [2.5 to 9.2] | 10.1 [4.8 to 21.1]
  Week 6 | 78.9 [49.9 to 124.8] | 100.3 [59.8 to 168.4] | 95.9 [54.6 to 168.3]
  Week 12 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 35.5 [19.6 to 64.5]
  Week 14 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 281.1 [166.6 to 474.1]
  Week 30/38 | 6.2 [2.6 to 14.8] | 11.5 [5.6 to 23.5] | 41.5 [22.6 to 75.9]
  Week 56/64 | 6.2 [2.5 to 15.4] | 10.6 [5.3 to 21.2] | 45.3 [26.0 to 79.0]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 4 = 0.823, 95% CI 2-sided [0.333 to 2.038]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 6 = 0.787, 95% CI 2-sided [0.410 to 1.508]
Statistical Analysis 3: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 30 = 0.535, 95% CI 2-sided [0.187 to 1.536]
Statistical Analysis 4: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; GMT Ratio (Group 1 / Group 2) at Week 56 = 0.590, 95% CI 2-sided [0.203 to 1.716]
Statistical Analysis 5: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 / Group 1) at Week 4 = 2.557, 95% CI 2-sided [0.972 to 6.731]
Statistical Analysis 6: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 / Group 1) at Week 6 = 1.215, 95% CI 2-sided [0.612 to 2.412]

14. Secondary Outcome: PRNT GMT 2 Weeks Following the Second Vaccination (Group 2 Compared to Group 1 and Group 3 (Combined))
Description: GMTs based on vaccinia-specific PRNT. Titers below the detection limit are included with a value of '1'.
Time Frame: Week 6
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 and 3 Combined | Group 2
Number analyzed (Participants) | 46 | 23
Titer | 88.1 [61.3 to 126.6] | 100.3 [59.8 to 168.4]
Statistical Analysis 1: Comparison: Group 1 and 3 Combined vs Group 2; Test type: Other; GMT Ratio (Group 1+3 [pooled] / Group 2) = 0.878, 95% CI 2-sided [0.480 to 1.606]

15. Secondary Outcome: PRNT GMT 2 Weeks Following the Last Vaccination
Description: GMTs based on vaccinia-specific PRNT. Titers below the detection limit are included with a value of '1'.
Time Frame: Week 6 (Groups 1 and 2), Week 14 (Group 3)
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
Titer | 78.9 [49.9 to 124.8] | 100.3 [59.8 to 168.4] | 281.1 [166.6 to 474.1]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT ratio (Group 1 [W6]/ Group 3 [W14) = 0.281, 95% CI 2-sided [0.146 to 0.542]
Statistical Analysis 2: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT ratio (Group 2 [W6]/ Group 3 [W14]) = 0.357, 95% CI 2-sided [0.178 to 0.718]

16. Secondary Outcome: PRNT GMT During Follow-up
Description: GMTs based on vaccinia-specific PRNT. Titers below the detection limit are included with a value of '1'. Participants discontinued prior to the follow-up visits are excluded.
Time Frame: Weeks 30 and 56 (Groups 1 and 2), Weeks 38 and 64 (Group 3)
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 18 | 22 | 24
Titer
  Week 30/38 | 6.2 [2.6 to 14.8] | 11.5 [5.6 to 23.5] | 41.5 [22.6 to 75.9]
  Week 56/64 | 6.2 [2.5 to 15.4] | 10.6 [5.3 to 21.2] | 45.3 [26.0 to 79.0]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 [W38]/ Group 1 [W30]) = 6.727, 95% CI 2-sided [2.493 to 18.150]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 3 [W64]/ Group 1 [W56]) = 7.275, 95% CI 2-sided [2.693 to 19.649]
Statistical Analysis 3: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 2 [W30]/ Group 3 [W38]) = 0.278, 95% CI 2-sided [0.115 to 0.672]
Statistical Analysis 4: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; GMT Ratio (Group 2 [W56]/ Group 3 [W64]) = 0.233, 95% CI 2-sided [0.100 to 0.541]

17. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: SC rate based on ELISA. SC is defined as the appearance of antibody titers >= detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 64 weeks
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
percentage of subjects
  Week 4 | 75.0 [50.9 to 91.3] | 82.6 [61.2 to 95.0] | 69.2 [48.2 to 85.7]
  Week 6 | 100.0 [83.2 to 100.0] | 100.0 [85.2 to 100.0] | 92.3 [74.9 to 99.1]
  Week 12 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 84.6 [65.1 to 95.6]
  Week 14 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 100.0 [86.8 to 100.0]
  Week 30/38: number analyzed (Participants) | 18 | 22 | 24
  Week 30/38 | 77.8 [52.4 to 93.6] | 72.7 [49.8 to 89.3] | 83.3 [62.6 to 95.3]
  Week 56/64: number analyzed (Participants) | 18 | 22 | 24
  Week 56/64 | 66.7 [41.0 to 86.7] | 68.2 [45.1 to 86.1] | 83.3 [62.6 to 95.3]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 4 = -7.6, 95% CI 2-sided [-34.1 to 17.9]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 6 = 0.0, 95% CI 2-sided [-16.8 to 16.3]
Statistical Analysis 3: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 30 = 5.1, 95% CI 2-sided [-24.5 to 32.6]
Statistical Analysis 4: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 56 = -1.5, 95% CI 2-sided [-31.5 to 29.2]
Statistical Analysis 5: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 3 - Gr 1) at Week 4 = -5.8, 95% CI 2-sided [-32.8 to 22.2]
Statistical Analysis 6: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 3 - Gr 1) at Week 6 = -7.7, 95% CI 2-sided [-25.1 to 10.1]

18. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA 2 Weeks Following the Second Vaccination (Group 2 Compared to Group 1 and Group 3 (Combined))
Description: as for outcome 17
Time Frame: Week 6
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 and 3 Combined | Group 2
Number analyzed (Participants) | 46 | 23
percentage of subjects | 95.7 [85.2 to 99.5] | 100.0 [85.2 to 100.0]
Statistical Analysis 1: Comparison: Group 1 and 3 Combined vs Group 2; Test type: Other; Difference in seroconversion rates (%) = -4.3, 95% CI 2-sided [-15.2 to 11.6]

19. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA 2 Weeks Following the Last Vaccination
Description: as for outcome 17
Time Frame: Week 6 (Groups 1 and 2), Week 14 (Group 3)
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
percentage of subjects | 100.0 [83.2 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [86.8 to 100.0]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 1 [W6] - Gr 3 [W14]) = 0.0, 95% CI 2-sided [-17.1 to 13.4]
Statistical Analysis 2: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 2 [W6] - Gr 3 [W14]) = 0.0, 95% CI 2-sided [-16.2 to 13.4]

20. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA During Follow-up
Description: as for outcome 17
Time Frame: Weeks 30 and 56 (Groups 1 and 2), Weeks 38 and 64 (Group 3)
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 18 | 22 | 24
percentage of subjects
  Week 30/38 | 77.8 [52.4 to 93.6] | 72.7 [49.8 to 89.3] | 83.3 [62.6 to 95.3]
  Week 56/64 | 66.7 [41.0 to 86.7] | 68.2 [45.1 to 86.1] | 83.3 [62.6 to 95.3]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr3 [W38] - Gr1 [W30]) = 5.6, 95% CI 2-sided [-19.6 to 33.0]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr3 [W64] - Gr1 [W56]) = 16.7, 95% CI 2-sided [-11.0 to 44.4]
Statistical Analysis 3: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr2 [W30] - Gr3 [W38]) = -10.6, 95% CI 2-sided [-35.6 to 14.3]
Statistical Analysis 4: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr2 [W56] - Gr3 [W64]) = -15.2, 95% CI 2-sided [-40.5 to 10.5]

21. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT
Description: SC rate based on PRNT. SC is defined as the appearance of antibody titers >= detection limit (2) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 64 weeks
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
percentage of subjects
  Week 4 | 60.0 [36.1 to 80.9] | 69.6 [47.1 to 86.8] | 80.8 [60.6 to 93.4]
  Week 6 | 100.0 [83.2 to 100.0] | 100.0 [85.2 to 100.0] | 96.2 [80.4 to 99.9]
  Week 12 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 96.2 [80.4 to 99.9]
  Week 14 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 1 | NA [NA to NA] — N/A=week 12 and 14 visits not scheduled for Group 2 | 100.0 [86.8 to 100.0]
  Week 30/38: number analyzed (Participants) | 18 | 22 | 24
  Week 30/38 | 72.2 [46.5 to 90.3] | 81.8 [59.7 to 94.8] | 91.7 [73.0 to 99.0]
  Week 56/64: number analyzed (Participants) | 18 | 22 | 24
  Week 56/64 | 66.7 [41.0 to 86.7] | 72.7 [49.8 to 89.3] | 95.8 [78.9 to 99.9]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 4 = -9.6, 95% CI 2-sided [-38.4 to 20.3]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 6 = 0.0, 95% CI 2-sided [-16.8 to 16.3]
Statistical Analysis 3: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 30 = -9.6, 95% CI 2-sided [-38.4 to 17.6]
Statistical Analysis 4: Comparison: Group 1 (Standard Regimen) vs Group 2 (Double Dose Regimen); Test type: Other; Diff in SC rate (Gr 1 - Gr 2) at Week 56 = -6.1, 95% CI 2-sided [-35.6 to 23.7]
Statistical Analysis 5: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 3 - Gr 1) at Week 4 = 20.8, 95% CI 2-sided [-7.7 to 47.8]
Statistical Analysis 6: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 3 - Gr 1) at Week 6 = -3.8, 95% CI 2-sided [-20.5 to 13.4]

22. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT 2 Weeks Following the Second Vaccination (Group 2 Compared to Group 1 and Group 3 (Combined))
Description: as for outcome 21
Time Frame: Week 6
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 and 3 Combined | Group 2
Number analyzed (Participants) | 46 | 23
percentage of subjects | 97.8 [88.5 to 99.9] | 100.0 [85.2 to 100.0]
Statistical Analysis 1: Comparison: Group 1 and 3 Combined vs Group 2; Test type: Other; Difference in seroconversion rates (%) = -2.2, 95% CI 2-sided [-12.0 to 13.2]

23. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT 2 Weeks Following the Last Vaccination
Description: as for outcome 21
Time Frame: Week 6 (Groups 1 and 2), Week 14 (Group 3)
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 20 | 23 | 26
percentage of subjects | 100.0 [83.2 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [86.8 to 100.0]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 1 [W6] - Gr 3 [W14]) = 0.0, 95% CI 2-sided [-17.1 to 13.4]
Statistical Analysis 2: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr 2 [W6] - Gr 3 [W14]) = 0.0, 95% CI 2-sided [-16.2 to 13.4]

24. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT During Follow-up
Description: as for outcome 21
Time Frame: Weeks 30 and 56 (Groups 1 and 2), Weeks 38 and 64 (Group 3)
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
Number analyzed (Participants) | 18 | 22 | 24
percentage of subjects
  Week 30/38 | 72.2 [46.5 to 90.3] | 81.8 [59.7 to 94.8] | 91.7 [73.0 to 99.0]
  Week 56/64 | 66.7 [41.0 to 86.7] | 72.7 [49.8 to 89.3] | 95.8 [78.9 to 99.9]
Statistical Analysis 1: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr3 [W38] - Gr1 [W30]) = 19.4, 95% CI 2-sided [-4.5 to 45.8]
Statistical Analysis 2: Comparison: Group 1 (Standard Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr3 [W64] - Gr1 [W56]) = 29.2, 95% CI 2-sided [5.8 to 55.4]
Statistical Analysis 3: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr2 [W30] - Gr3 [W38]) = -9.8, 95% CI 2-sided [-33.0 to 11.7]
Statistical Analysis 4: Comparison: Group 2 (Double Dose Regimen) vs Group 3 (Booster Regimen); Test type: Other; Diff in SC rate (Gr2 [W56] - Gr3 [W64]) = -23.1, 95% CI 2-sided [-46.7 to -1.0]

ADVERSE EVENTS:
Time Frame: within 75 weeks
Arm/Group | Group 1 (Standard Regimen) | Group 2 (Double Dose Regimen) | Group 3 (Booster Regimen)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 2/31
Other Adverse Events (participants affected / at risk) | 5/27 | 6/29 | 10/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Standard Regimen) (N=27) | Group 2 (Double Dose Regimen) (N=29) | Group 3 (Booster Regimen) (N=31)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Standard Regimen) (N=27) | Group 2 (Double Dose Regimen) (N=29) | Group 3 (Booster Regimen) (N=31)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-11-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT02038881/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT02038881/SAP_001.pdf